CLINICAL TRIAL: NCT02093572
Title: Effect of Skipping Breakfast on Metabolic Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201402039; KL2TR000450 (NIH)
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Skipping Breakfast; Circadian Rhythms
Keywords: Clock genes; Metabolism; Insulin sensitivity
MeSH Terms: conditions — Intermittent Fasting; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Experimental): Subjects randomized to this group will consume 3 standard meals/day during the 2 week intervention period of the study.
  Interventions: Other: 3 standard meals/day
- Breakfast skipping (Experimental): Subjects randomized to this group will consume 2 meals/day (omit breakfast - with caloric intake equal to consuming 3 meals/day) during the 2 week intervention period of the study.
  Interventions: Other: 2 meals/day (omit breakfast)

INTERVENTIONS:
Other: 3 standard meals/day
  Arms: Control
Other: 2 meals/day (omit breakfast)
  Arms: Breakfast skipping

SUMMARY:
The purpose of this study is to test the hypothesis that the disruption of the "normal" (three meals a day) eating pattern and prolonged overnight fasting caused by skipping breakfast: i) alters the expression of specific clock genes and clock gene targets involved in regulating adipose tissue lipolysis (breakdown or destruction); ii) increases basal adipose tissue lipolytic (breakdown) activity and plasma free fatty acid (FFA) concentrations; iii) reduces skeletal muscle insulin sensitivity; and iv) increases daylong plasma glucose, FFA, and insulin concentrations. The investigator will do this by studying healthy, lean persons either randomized to consume either 3 standard meals per day or omit breakfast and consume 2 meals per day without changing daily calorie intake (skipping breakfast group).

ELIGIBILITY:
Inclusion Criteria:

* Males & females
* 18-55 years old
* BMI between 18.5 - 29.9 kg/m²
* Sleeps >7 hours/night
* Normally consume 3 meals/day, including breakfast

Exclusion Criteria:

* Pregnancy, lactating or breastfeeding
* Diabetes
* Sleep disorders
* Significant organ dysfunction
* Shift or nighttime workers
* Smokers
* Breakfast skippers
* People who regularly sleep <7 hours/night
* Consume excess amounts of alcohol
* Medications that could alter the results of this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Determine the effect of skipping breakfast on basal adipose tissue lipolytic activity and skeletal muscle insulin sensitivity | 3 weeks
  Hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotopically labeled trace infusions will be conducted before and after the diet intervention to asses the changes on basal adipose tissue lipolytic activity and skeletal muscle insulin sensitivity.
Determine the effect of skipping breakfast on 24-hour plasma substrate, hormone concentrations and intramyocellular fatty acid mediators of lipotoxicity. | 3 weeks
  Multiple blood and skeletal muscle biopsy samples will be obtained during a 24-hour feeding study before and after the diet intervention to assess 24-hour plasma substrate, hormone concentrations and intramyocellular fatty acid mediators of lipotoxicity.
Determine the effect of skipping breakfast on the diurnal expression of clock genes and downstream metabolic targets involved in regulating adipose tissue lipolytic activity and skeletal muscle insulin action. | 3 weeks
  Serial biopsy samples (every 6 hours) of adipose tissue and muscle will be obtained during the 24-hour feeding study to evaluate diurnal expression patterns of i) clock genes [CLOCK, brain and muscle Arnt-like protein-1(BMAL1), period1 (PER1), period2 (PER2), and Dbp D site albumin promoter binding protein (DBP)] in adipose tissue and muscle and ii) putative downstream clock gene targets associated with lypolysis in adipose tissue [hormone-sensitive lipase(HSL) and adipocyte triglyceride lipase (ATGL)], skeletal muscle insulin action [glucose transporter type 4(GLUT4)] and skeletal muscle fatty acid metabolism [cluster of differentiation 36(CD36), uncoupling protein 3 (UCP3) and pyruvate dehydrogenase kinase, isozyme 4(PDK4)].

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yoshino, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Yamaguchi S, Moseley AC, Almeda-Valdes P, Stromsdorfer KL, Franczyk MP, Okunade AL, Patterson BW, Klein S, Yoshino J. Diurnal Variation in PDK4 Expression Is Associated With Plasma Free Fatty Acid Availability in People. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1068-1076. doi: 10.1210/jc.2017-02230. PMID 29294006